CLINICAL TRIAL: NCT05474625
Title: Efficacy of High-intensity Laser Therapy (HILT) in the Patients With Cervical Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Şükran Güzel, Asst. Prof., Baskent University Ankara Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-946003339-604.01.02-38865
Record Dates: First submitted 2022-07-13; First posted 2022-07-26 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Cervical Disc Herniation
MeSH Terms: interventions — Ultrasonography; Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise Group (Active Comparator): Only exercises
  Interventions: Other: Exercise
- High Intensity Laser Therapy(HILT) Group (Active Comparator): Exercises+HILT
  Interventions: Device: High Intensity Laser Therapy; Other: Exercise
- Conventional Physiotherapy Group (Active Comparator): Exercise+Hotpack+Transcutaneous nerve stimulation (TENS)+Ultrasound
  Interventions: Device: Ultrasound; Device: Transcutaneous nerve stimulation (TENS); Other: Exercise

INTERVENTIONS:
Device: High Intensity Laser Therapy — For each 25 cm² of painful area, 1.02 minutes of treatment will give in the analgesic phase, with an energy of 8.0 watt, a dose of 5 Joules/ cm², a frequency of 25 Hertz(Hz) and a total energy of 125 joules. The application time for one session was approximately 15 minutes. Total 15 sessions will be applied to the neck area for a period of 3 weeks, 5 days a week.
  Arms: High Intensity Laser Therapy(HILT) Group
Device: Ultrasound — This treatment was applied to the cervical paravertebral region with a direct contact with the skin with the aid of an ultrasonic gel, at a dose of 1 megahertz(MHz) and 1.5 Watt/cm² for 4 minutes
  Arms: Conventional Physiotherapy Group
Device: Transcutaneous nerve stimulation (TENS) — TENS was performed using 4 adhesive electrodes 5 × 5 cm size in the cervical paravertebral region, 80 Hertz (Hz) frequency and 180 miliseconds current for 20 minutes.
  Arms: Conventional Physiotherapy Group
Other: Exercise — A specific program consisted of 15 minutes exercise sessions was provided under the supervision of a physiotherapist . All patients will perform isometric strengthening exercises, active range of motion exercises, and cervical region stretching exercises for 15 sessions (during 3 weeks, on weekdays).

SUMMARY:
The worldwide prevalence of neck pain is between 16.7-75.1%, it has been seen at an increasing rate in recent years due to sedentary living conditions.

Pharmacological treatment, neck collar, traction, manual therapy, interventional injection techniques, surgical treatment and conventional physical therapy methods such as hotpack, ultrasound, TENS (Transcutaneous electrical nerve stimulation), vacuum interference, exercise are applied in the treatment of neck pain.

In recent years, High Intensity Laser Therapy (HILT) has been used as a painless and non-invasive physical therapy agent. It received FDA approval in 2002 for HILT in the treatment of variety of musculoskeletal disorders.

There are a few studies in the literature investigating the efficacy of HILT in chronic neck pain. There is only one study investigating the efficacy of HILT in cervical disc herniation. In this study, the efficacy of HILT and ultrasound-TENS in the treatment of neck pain caused by cervical disc herniation has been compared, but the results of the exercise control group and long-term follow-up were not available.

The aim of this randomized controlled trial is to evaluate the short and long-term efficacy of HILT treatment using improvement in the pain, range of motion, activities of daily living and functionality of the cervical spine in patients with cervical disc herniation. In group 1, only exercises will be applied; in the group 2, HILT will be applied in addition to exercise; in the group 3, hotpack, TENS, ultrasound will be applied in addition to exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical disc herniation diagnosed by MRI whose symptoms started for at least 3 months ago
* Not receiving physical therapy and rehabilitation in the last 3 months
* Not taking any medications such as analgesics, anti-inflammatoires or muscle relaxants for the treatment of symptoms.

Exclusion Criteria:

* patients with major psychiatric disease, cervical spine surgery and rheumatological disease; pacemaker users; those who were injected with local corticosteroids; pregnant women; cancer patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | Pre-treatment
  This scale is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Scoring was between 0-50, where high scores indicate a poor result
Neck Disability Index | 1. month
  This scale is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Scoring was between 0-50, where high scores indicate a poor result
Neck Disability Index | 3. month
  This scale is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Scoring was between 0-50, where high scores indicate a poor result

SECONDARY OUTCOMES:
Short Form Health Survey-36 | pre-treatment
  A generic health survey which assesses health concepts that are pertinent to functional status and well-being such as physical function, bodily pain, role limitation due to emotional and physical problems. The sub scale values are reported: physical functioning, bodily pain, vitality, general health, social functioning, role limitation due to emotional problems, role limitation due to physical problems, mental health. The lowest and highest possible raw score for the subscales are as follows: physical functioning 10-30, physical role 4- 8, bodily pain 2-12, general health 5-25, vitality 4-24, social functioning 2-10, emotional role 3-6, mental health 5-30. Higher values signify better well being in all subgroups. The raw score is then used to calculate the 'transformed scale: Transformed scale= [(actual raw score- lowest possible raw score)/possible raw score range]100.
Short Form Health Survey-36 | 1. months
  A generic health survey which assesses health concepts that are pertinent to functional status and well-being such as physical function, bodily pain, role limitation due to emotional and physical problems. The sub scale values are reported: physical functioning, bodily pain, vitality, general health, social functioning, role limitation due to emotional problems, role limitation due to physical problems, mental health. The lowest and highest possible raw score for the subscales are as follows: physical functioning 10-30, physical role 4- 8, bodily pain 2-12, general health 5-25, vitality 4-24, social functioning 2-10, emotional role 3-6, mental health 5-30. Higher values signify better well being in all subgroups. The raw score is then used to calculate the 'transformed scale: Transformed scale= [(actual raw score- lowest possible raw score)/possible raw score range]100.
Short Form Health Survey-36 | 3. months
  A generic health survey which assesses health concepts that are pertinent to functional status and well-being such as physical function, bodily pain, role limitation due to emotional and physical problems. The sub scale values are reported: physical functioning, bodily pain, vitality, general health, social functioning, role limitation due to emotional problems, role limitation due to physical problems, mental health. The lowest and highest possible raw score for the subscales are as follows: physical functioning 10-30, physical role 4- 8, bodily pain 2-12, general health 5-25, vitality 4-24, social functioning 2-10, emotional role 3-6, mental health 5-30. Higher values signify better well being in all subgroups. The raw score is then used to calculate the 'transformed scale: Transformed scale= [(actual raw score- lowest possible raw score)/possible raw score range]100.
Visual Analog Scale | pre-treatment
  The Visual Analog Scale provides a subjective, visual linear pain score from 0 to 10 cm scored by the patient where 0 cm is no pain.
Visual Analog Scale | 1. month
  The Visual Analog Scale provides a subjective, visual linear pain score from 0 to 10 cm scored by the patient where 0 cm is no pain.
Visual Analog Scale | 3. month
  The Visual Analog Scale provides a subjective, visual linear pain score from 0 to 10 cm scored by the patient where 0 cm is no pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Ankara Hospital, Ankara, Turkey (Türkiye)